CLINICAL TRIAL: NCT05287945
Title: A Phase I/II, Open-Label, Single-Arm Study on Safety, Tolerability and Anti-Tumour Efficacy of Orellanine Treatment in Patients With Metastatic Clear-Cell or Papillary Renal Cell Carcinoma
Brief Title: Study of Orellanine in Metastatic Clear-Cell or Papillary Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncorena AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC001-CL-001
Record Dates: First submitted 2021-05-24; First posted 2022-03-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — orellanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orellanine (Experimental): Orellanine administered intravenously
  Interventions: Drug: Orellanine

INTERVENTIONS:
Drug: Orellanine — Orellanine administered intravenously

SUMMARY:
A phase I/II, open-label, study to determine the safety and preliminary efficacy of orellanine in patients with metastatic clear-cell or papillary renal carcinoma.

DETAILED DESCRIPTION:
This is an open, non-controlled, phase I/II study evaluating the safety, tolerability, and anti-tumor efficacy of orellanine treatment in patients with metastatic clear-cell or papillary renal carcinoma. The study will include up to 75 patients. The phase I will consist of 3 parts: Part A - an intra-patient dose escalation part, followed by a dose exposure (Part B), followed by a dose expansion (Part C).

ELIGIBILITY:
Inclusion criteria:

1. Has provided written informed consent.
2. Has a diagnosis of histologically confirmed advanced ccRCC or pRCC. No conventional therapy is available or considered appropriate by the treating physician or is declined by the patient.
3. For patients in the expansion portion of the study only: Measurable disease per RECIST version 1.1 criteria.
4. ECOG performance status of 0 - 2.
5. Age ≥18 years.
6. Life expectancy ≥3 months.
7. Has acceptable haematologic laboratory values defined as:

   1. Neutrophils ≥1.5 × 10^9/L, without growth factor stimulation within 3 weeks prior to the blood test;
   2. Platelets ≥100 × 10^9/L;
   3. Haemoglobin ≥5.6 mmol/L (~90 g/L). Use of erythropoietin or blood transfusions are permitted.
8. Has acceptable liver laboratory values defined as:

   1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN (≤5 × ULN for patients with liver metastases
   2. Total bilirubin ≤1.5 × ULN or direct bilirubin ≤ ULN for patients with total bilirubin levels >1.5 × ULN
   3. For patients diagnosed with Gilbert's syndrome, total bilirubin ≤2 × ULN is acceptable.
9. Must be on chronic hemodialysis (on a consistent regimen for the previous three months, with allowance for intermittent treatments as required for volume overload).
10. The patient's treating nephrologist and oncologist agree that the prospect of loss of remaining renal function resulting from this treatment will not significantly change the patient's future and chronic dialysis treatment.
11. Female patients of child-bearing potential and male patients must agree to use 2 forms of highly effective contraception for the duration of study treatment and after the last dose of orellanine for at least 3 months for males and 6 months for females.
12. For females of child-bearing potential, a negative serum pregnancy test at screening.
13. Patients who are willing and able to comply with travel requirements, scheduled visits, treatment schedule, efficacy assessments, laboratory tests, and other study procedures.

Exclusion criteria:

1. Diagnosis of any other malignancy within 2 years prior to enrolment, except for adequately treated basal cell or squamous cell skin cancer, superficial melanoma, or carcinoma in situ of the breast or of the cervix, or low grade (Gleason 7 or below) prostate cancer on surveillance with no plans for treatment intervention (e.g., surgery, radiation, or castration)
2. Radiotherapy within 2 weeks before first dose.
3. Immuno-oncology therapy (IO) given in the last six (6) months prior to enrolment
4. Other systemic anti-cancer therapy within 2 weeks before first dose.
5. Has not recovered from AEs due to prior anti-cancer medications to at least grade 1 by CTCAE version 5.0 (except for alopecia and grade 2 neuropathy).
6. Has received any other investigational product within 4 weeks before first dose.
7. Pregnant or breastfeeding women.
8. Uncontrolled medical condition including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements, or would, in the opinion of the investigator, place the patient at increased risk.
9. QTc interval at baseline of ≥470 msec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Adverse events and laboratory abnormalities as graded by NCI CTCAE v5.0. | Through study completion, approximately 1 year
Changes in arterial blood pressure measurements | Through study completion, approximately 1 year
Changes in pulse rate measurements | Through study completion, approximately 1 year
Changes in respiratory rate measurements | Through study completion, approximately 1 year
Changes in temperature measurements | Through study completion, approximately 1 year
Changes in physical examination findings | Through study completion, approximately 1 year
Maximum tolerable dose of orellanine | Through study completion, approximately 1 year

SECONDARY OUTCOMES:
Efficacy of orellanine based on time to tumor response | Through study completion, approximately 1 year.
Efficacy of orellanine based on best overall response | Through study completion, approximately 1 year.
Area under the curve extrapolated to infinity | Through study completion, approximately 1 year.
Terminal half-life | Through study completion, approximately 1 year.
Partial area under the curve | Through study completion, approximately 1 year.
Dose proportionality | Through study completion, approximately 1 year.
Time to maximum plasma concentration | Through study completion, approximately 1 year.
Maximum plasma concentration | Through study completion, approximately 1 year.
Total body clearance | Through study completion, approximately 1 year.
Volume of distribution | Through study completion, approximately 1 year.

CONTACTS AND LOCATIONS:
Locations (2):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Pursuant to relevant data protection and privacy legislation, patients will authorize the collection, use and disclosure of their study data by the investigator and by those persons who need that information for the purposes of the study.

REFERENCES:
- [Background] Buvall L, Hedman H, Khramova A, Najar D, Bergwall L, Ebefors K, Sihlbom C, Lundstam S, Herrmann A, Wallentin H, Roos E, Nilsson UA, Johansson M, Tornell J, Haraldsson B, Nystrom J. Orellanine specifically targets renal clear cell carcinoma. Oncotarget. 2017 Jul 25;8(53):91085-91098. doi: 10.18632/oncotarget.19555. eCollection 2017 Oct 31. PMID 29207627
- [Background] Dy GW, Gore JL, Forouzanfar MH, Naghavi M, Fitzmaurice C. Global Burden of Urologic Cancers, 1990-2013. Eur Urol. 2017 Mar;71(3):437-446. doi: 10.1016/j.eururo.2016.10.008. Epub 2016 Oct 28. PMID 28029399
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Hedman H, Holmdahl J, Molne J, Ebefors K, Haraldsson B, Nystrom J. Long-term clinical outcome for patients poisoned by the fungal nephrotoxin orellanine. BMC Nephrol. 2017 Apr 3;18(1):121. doi: 10.1186/s12882-017-0533-6. PMID 28372584
- [Background] Merza H, Bilusic M. Current Management Strategy for Metastatic Renal Cell Carcinoma and Future Directions. Curr Oncol Rep. 2017 Apr;19(4):27. doi: 10.1007/s11912-017-0583-8. PMID 28303494
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949